CLINICAL TRIAL: NCT04689594
Title: A Phase III, Multicenter, Open-label Study to Evaluate the Esophageal Stenosis Inhibition Effects and Safety of CLS2702C/CLS2702D After Endoscopic Submucosal Dissection (ESD) in Patients With Superficial Esophageal Cancer in the Steroid Administration Risk Group
Brief Title: A Study to Evaluate the Esophageal Stenosis Inhibition Effects of CLS2702C/CLS2702D After Endoscopic Submucosal Dissection (ESD) in Patients With Superficial Esophageal Cancer in the Steroid Administration Risk Group
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the extension of the clinical trial period due to a problem that occurred in the first patient of this study, there were concerns about business viability, so we decided to cancel this study.
Sponsor: CellSeed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLS2702-ESO-02
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Superficial Esophageal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLS2702C/CLS2702D (Experimental)
  Interventions: Combination Product: CLS2702C/CLS2702D

INTERVENTIONS:
Combination Product: CLS2702C/CLS2702D — CLS2702C (cell sheet) will be transplanted to the wound site using CLS2702D (transplantation device) (screening period, 1 month [4 weeks]; cell sheet culture period, 0.5 month; transplantation and assessment period, 6 months [24 weeks]); follow-up period, 6 months [24 weeks]) Other Names: •Human (autologous) oral mucosal cell sheet
  •Transplantation device

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of esophageal epithelial regenerative treatment by the transplantation of the product, CLS2702C, to the esophageal wound site after extensive ESD for superficial esophageal cancer in the steroid administration risk group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to undergo ESD for the treatment of superficial esophageal cancer
2. Patients aged >=20 years at the time of consent
3. Patients with no clinical metastasis (cN0M0) by cervical to abdominal CT
4. Patients with an endoscopically diagnosed depth of wall invasion remaining in the epithelium (EP) or lamina propria mucosae (LPM)
5. Patients with a tumor diagnosed as >=50% and <100% of circumference, and with prediction that resection circumference will be >=75% and <100%.
6. Patients with a tumor the major axis is <=50 mm, and with prediction that a major axis of a resection will be <=80 mm.
7. If the patient has multiple lesions, the circumference of all minor lesions other than the one lesion with the largest circumference (major lesion) must be <50%. However, if it is predicted that the major axis of the mucosal defect is >80 mm due to treating the major and minor lesions and assembling ulcers after the treating, the patient is excluded.
8. Patients with squamous cell carcinoma (including high-grade intraepithelial neoplasia) as confirmed by biopsy
9. Patients whose lesion is confirmed to be localized in the thoracic esophagus (lesions in the cervical esophagus or abdominal esophagus will be excluded). The location of the lesion will be determined by endoscopy.
10. Patients who have not received pretreatment for esophageal cancer. Treatment by ESD for superficial esophageal cancer for which the depth of wall invasion has been assessed to remain in the epithelium (EP) or lamina propria mucosae (LPM) is not included in the definition of pretreatment. However, patients who have a scar due to previous ESD in the major or minor lesions will be excluded from the study.
11. Patients with an ECOG Performance Status (PS) of 0 or 1
12. Patients in whom a commonly used endoscope with a tip diameter of 8.9 mm can pass
13. Patients with a dysphagia score of 0
14. Patients whose laboratory values within 28 days before enrolment meet all of the following criteria:

    * White blood cell count: >=4,000/microL
    * Platelet count: >=100,000/microL
    * AST: <=100 IU/L
    * ALT: <=100 IU/L
    * Total bilirubin: <=2.0 mg/dL
    * Serum creatinine: <=2.0 mg/dL
15. Patients who have received sufficient explanation about the study and provided written voluntary consent.
16. Patients who meet any of the following criteria:

    * With fibrous nodule shadow on IGRA negative diagnostic imaging
    * Required continuous systemic administration of immunosuppressants
    * With diabetes with blood glucose level of 180 mg/dL or more 2 hours after meal even with insulin
    * With 7.0% or more of hemoglobin A1c (HbA1c, (International standard value (NGSP value)) even if taking 2 or more drug treatments for more than 3 months
    * With high blood pressure which does not reach the target value even if taking 2-3 antihypertensive drugs or reach it with 4 or more antihypertensive drugs
    * With glaucoma, posterior capsule cataract or herpes simplex keratitis (Ophthalmology consultation is not mandatory)
    * With a risk of administration of corticosteroids based on medical judgment.

Exclusion Criteria:

1. Patients with cardiac disease (myocardial infarction, unstable angina, and heart failure), renal disease (nephrotic syndrome and kidney failure)
2. Patients who have an active (within 1 year) malignancy other than esophageal cancer
3. Patients with active bacterial, fungal, or viral infection
4. Patients who are being treated with a corticosteroid except for topical corticosteroids (ointments and creams) and oral ointments or patches used for treating stomatitis after oral mucosal tissue taken from D-16 to D-1.
5. Patients who are positive for any of serological test (HBs antigen, HBc antibody/HBs antibody, HCV antibody, HIV-1/2 antibody, HTLV-1 antibody, syphilis treponema antibody) or nucleic acid amplification test (HBV-DNA, HCV-RNA, HIV-RNA). However, this does not apply if the HBs antibody is positive and HBV-DNA is negative and the reason is clear that he was vaccinated with the hepatitis B vaccine.
6. Patients with a mental disorder that is difficult to control
7. Pregnant women, lactating women, and potentially pregnant women
8. Patients who have participated in another clinical study within 6 months, those who are participating in another clinical study, and those who plan to participate in another clinical study during participation in this study
9. Patients from whom tissues cannot be collected due to a disease (e.g., stomatitis, erosion, mass, and blister) in the oral mucosa at the tissue collection site
10. Patients with a history of hypersensitivity to antibiotic preparations (ampicillin sodium, sulbactam sodium, streptomycin sulfate, gentamicin sulfate, or amphotericin B) or who have taken drugs that may affect the study (within 28 days before enrolment)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects without stenosis | 24 weeks after endoscopic
  Proportion of participants without stenosis until 24 weeks after endoscopic submucosal dissection (ESD)

CONTACTS AND LOCATIONS:
Locations (1):
- Okayama University Hospital, Okayama, Japan